CLINICAL TRIAL: NCT05615766
Title: EXO4UL- Assessment of a Robotic Exoskeleton for Upper Limb Rehabilitation of Spinal Cord Injured Patients
Brief Title: Assessment of a Robotic Exoskeleton for Upper Limb Rehabilitation
Acronym: Exo4UL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government); The Queen Elizabeth National Spinal Injuries Unit, Scotland (Unknown); Stoke Mandeville Spinal Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRAS312522
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Device Intervention (Experimental): The intervention group who will be undergoing rehabilitation using the robotic exoskeleton in addition to the assigned traditional rehabilitation programme on their dominant arm only.
  Interventions: Device: Experimental: Device Intervention
- Control (No Intervention): the matched control group will be the same subjects undergoing traditional rehabilitation only on their non-dominant arm.

INTERVENTIONS:
Device: Experimental: Device Intervention — The robotic rehabilitation programme using the MARK from Myomo (myomo.com) for the intervention group will last for 12 weeks with up to four sessions of rehabilitation per week, i.e. total of 48 sessions. Spinal cord injured inpatients in the study will have this intervention on their dominant arm in addition to the traditional rehabilitation programme assigned and standard care.
  Other Names: Robotic Rehabilitation
  Arms: Device Intervention

SUMMARY:
Rehabilitation robotics has the potential to facilitate rehabilitation at home and empower people with spinal injuries to self-manage increasing their independence and improving their quality of life.

The objective of this study is to assess for the first time in the NHS the efficacy of a commercial robotic orthosis for upper limb rehabilitation in patients with spinal cord injury. The device is produced by Myomo (myomo.com) which is an American company. We will be assessing the wearable robotic orthosis also known as robotic exoskeleton in two different neuro-rehabilitation centres: National Spinal injuries Unit in Glasgow (Scotland) and The Robert Jones and Agnus Hunt Orthopaedic Hospital in Oswestry (England). The study will involve nine spinal cord injured tetraplegic inpatients in total.

Patients will follow a twelve-week rehabilitation programme with three to four sessions per week in addition to their usual care and rehabilitation. Each session lasts for approximately 45 minutes. Participants arm function, range of motion, spasticity level will be measured before, half-way and at the end of the programme to assess change in these and other parameters. Training will focus on the dominant arm of the patient and compared to the other arm at every assessment stage.

We shall evaluate therapists' and patients' satisfaction with the commercial device in addition to assessing various clinical measures to evaluate the efficacy of using the robotic orthosis in rehabilitation and recovery of arm function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years.
* The levels of C5 C6 Asia C/D would provide individuals with elbow and hand impairment and potentially functional shoulder movements. C7, C8 individuals could also benefit from the hand component of the device.
* Some gross shoulder movement at start of the trial to enable changes at the elbow/hand, to have the greatest potential for functional change.
* Preservation of hand sensation as base for motor restoration.
* Some sitting balance would give the best opportunity for the arm to be released for functional upper limb activity.
* EMG (muscle activity) evidence of active finger flexion, extension and elbow flexion extension Grade 1-2.
* Minimal or No community functional use of upper limb at start of trial.
* Spasticity MAS 1-3/5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Independence Measure version III (SCIM III) | Change from baseline (week 1) at 6 weeks
  assesses performance in activities of daily living and mobility for individuals with spinal cord injury
Spinal Cord Independence Measure version III (SCIM III) | Change from baseline (week 1) at 12 weeks
  assesses performance in activities of daily living and mobility for individuals with spinal cord injury

SECONDARY OUTCOMES:
The Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP). | Change from baseline (week 1) at 6 weeks and 12 weeks
  The GRASSP is a clinical impairment measure for the upper limb for use after tetraplegia. The measure includes three domains which are important in describing hand function.
The modified Ashworth scale | Change from baseline (week 1) at 6 weeks and 12 weeks
  Ashworth scale is the most universally accepted clinical spasticity assessment tool used to measure the increase of muscle tone.
Range of Motion | Change from baseline (week 1) at 6 weeks and 12 weeks
  to assess the capability of a joint to go through its complete spectrum of movements
Canadian Occupational Performance Measure (COPM) | Change from baseline (week 1) at 6 weeks and 12 weeks
  COPM assesses the patient's perceived occupational performance in the areas of selfcare, productivity, and leisure

OTHER OUTCOMES:
The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | Change from baseline (week 1) at 6 weeks and 12 weeks
  The QUEST 2.0 evaluates a patient's satisfaction with various assistive technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Lakany, PhD, Principal Investigator — University of Liverpool; Simon J Pickard, Study Director — Robert Jones and Agnes Hunt Orthopaedic Hospital
Locations (2):
- United Kingdom (2):
  - Royal National Orthopaedic Hospital (Stanmore), London
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry